CLINICAL TRIAL: NCT05697393
Title: External Upper Esophageal Sphincter Band (Shaker Pressure Band) and Gastroesophageal Reflux Disease
Brief Title: External UES Band (Shaker Pressure Band) and GERD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, Reza Shaker, MD, Associate Provost for Clinical and Translational Research, Senior Associate Dean and Director of the Clinical and Translational Science Institute of SE WI, and the Joseph E. Geenen Professor and Chief of Gastroenterology and Hepatology, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO00014424
Record Dates: First submitted 2023-01-13; First posted 2023-01-25 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (2):
- Shaker Pressure Band GERD patients with external laryngeal pressure (Active Comparator): One week of Shaker pressure band
  Interventions: Device: Shaker Pressure Band
- Shaker Pressure Band GERD patients without external laryngeal pressure (Placebo Comparator): One week of sham Shaker pressure band (no external laryngeal pressure)
  Interventions: Device: Shaker Pressure Band

INTERVENTIONS:
Device: Shaker Pressure Band

SUMMARY:
This protocol is a study to assess the efficacy of an external upper esophageal band to decrease subjective nighttime symptoms related to esophageal reflux into the pharynx.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease is the most common malady of the esophagus. It is estimated that 7-10% of the US population suffers from various degrees of this disease. This translates into a significant burden on health care resources. However, complications of reflux disease induced outside the esophagus; namely in the aerodigestive and airway tracts, are only recently becoming more recognized. For example, it is estimated that 4-10% of laryngeal diseases seen in ear, nose and throat clinics are associated with reflux disease. Although these supra-esophageal complications have become recognized as significant clinical problems, until recently the physiology and pathophysiology of interactions between the esophagopharyngeal and pharyngo-laryngeal axes during retrograde transit through the esophagus and pharynx had remained for the most part unexplored. In-depth investigation of this functional relationship and the mechanisms that prevent retrograde aspiration is of significant clinical importance not only because of pharyngo-laryngeal complications of reflux, but because of the devastating consequences of retrograde aspiration into the lungs and its complications, such as pneumonia, pneumonitis, lung fibrosis and abscesses, especially in the senior citizen group. Although much has been learned about the mechanism of airway protection against reflux of gastric content into the pharynx and larynx, during the last funding period there remains a substantial gap in our knowledge in this field, many questions remain unanswered. The progress achieved previously has provided the necessary basis to close some of these fundamental gaps in our knowledge through the hypotheses driven studies proposed.

The investigators know that patients can have significant gastroesophageal reflux during the sleeping state despite maximum medical therapy and lifestyle modifications. These patients experience severe nighttime and daytime symptoms that can have significant effect on their overall health. The investigators are proposing a non-invasive approach to help decrease reflux events beyond the upper esophageal sphincter.

Esophageal reflux into the pharynx can cause persistent symptoms such as severe heartburn, chest pain, voice hoarseness, cough, choking and sleep disturbances. There is evidence that external pressure to the upper esophageal sphincter can decrease the amount of reflux into the pharynx and possibly decrease these subjective symptoms. The investigators have anecdotal clinical evidence that an external band placed at the level of the cricoid cartilage can alleviate these symptoms in a carefully selected cohort of patients with true reflux into their pharynx. It is postulated that this external band can increase the luminal pressure at the upper esophageal sphincter (UES) and thus decrease esophageal reflux into the pharynx. The external band is titrated to an internal pressure of 20 mmHg. This measurement is based on preliminary data and previous studies that have shown that a driving reflux pressure is equal to or greater than 20 mmHg.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be 18 years of age or older.
* Patients with gastroesophageal reflux disease (GERD) who has ear, nose, and throat symptoms, chronic cough, choking, or regurgitation (food coming back up into the throat).
* The patient has been diagnosed with GERD with extra-esophageal symptoms, esophagitis, hiatal hernia, achalasia, or diffuse esophageal spasm.
* The patient must not be pregnant or lactating.

Exclusion Criteria:

* The patient cannot be younger than 18 years of age or older than 85.
* The patient cannot have sleep apnea or be on CPAP
* Patient cannot have previous head or neck surgery or radiation.
* Patient cannot have carotid artery disease, thyroid disease or history of cerebral vascular disease.
* Patients with an inability to tolerate nasal intubation.
* Patients with significant bleeding disorders for whom nasal intubation has been deemed contraindicated
* Patients with a known esophageal obstruction prevent passage of the manometry probe.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2011-01-25 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Symptom Analysis | Initial physician assessment and after one week of treatment
  Patients will be evaluated and categorized by their symptoms at the time of their clinical physician's assessment. All patients will then undergo the same study procedures already approved for this protocol and evaluate the change in their symptoms using the evaluation forms currently available in this protocol.

CONTACTS AND LOCATIONS:
Overall Officials: Reza Shaker, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No